CLINICAL TRIAL: NCT03439072
Title: G-Pen™ (Glucagon Injection) Compared to Lilly Glucagon (Glucagon for Injection [RDNA Origin]) for Induced Hypoglycemia Rescue in Adults With T1D: a Phase 3 B Multi-Centered, Randomized, Controlled, Single Blind, 2-Way Crossover Study to Evaluate Efficacy and Safety
Brief Title: G-Pen™ Compared to Lilly Glucagon for Hypoglycemia Rescue in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Collaborators: SGS S.A. (Industry); Integrated Medical Development (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: XSGP-303
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Results first posted 2019-05-30 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Insulin Hypoglycemia; Type 1 Diabetes Mellitus; Severe Hypoglycemia
Keywords: glucagon; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- G-Pen followed by Lilly Glucagon (Other): 1 mg G-Pen at the first treatment visit followed by 1 mg Lilly Glucagon at the second treatment visit
  Interventions: Drug: G-Pen; Drug: Lilly Glucagon
- Lilly Glucagon followed by G-Pen (Other): 1 mg Lilly Glucagon at the first treatment visit followed by 1 mg G-Pen at the second treatment visit
  Interventions: Drug: G-Pen; Drug: Lilly Glucagon

INTERVENTIONS:
Drug: G-Pen — 1 mg subcutaneous injection of G-Pen (glucagon injection) administered via auto-injector
  Other Names: glucagon
Drug: Lilly Glucagon — 1 mg subcutaneous injection of Lilly Glucagon (glucagon injection [RNDA Origin])
  Other Names: GEK

SUMMARY:
This is a non-inferiority, multi-center, randomized, controlled, single-blind, two-way crossover efficacy and safety study in subjects with Type 1 diabetes mellitus. The study involves two daytime clinical research center (CRC) visits with random assignment to receive G-Pen™ glucagon 1 mg during one period and Lilly Glucagon 1 mg during the other. Each daytime visit is preceded by an overnight stay in the CRC. In the morning of the inpatient study visit, the subject is brought into a state of hypoglycemia through IV administration of regular insulin diluted in normal saline. After a hypoglycemic state with plasma glucose < 50 mg/dL is verified, the subject is administered a dose of G-Pen or Lilly Glucagon via subcutaneous injection. Plasma glucose levels are monitored for up to 180 minutes post-dosing, with a value of >70.0 mg/dL within 30 minutes of glucagon administration indicating a positive response. After 3 hours, the subject is given a meal and discharged when medically stable. After a wash-out period of 7 to 28 days, subjects return to the CRC, and the procedure are repeated with each subject crossed over to the other treatment. A follow-up visit as a safety check is conducted 2-7 days following administration of the final dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females diagnosed with type 1 diabetes mellitus for at least 24 months.
2. Current usage of daily insulin treatment that includes having an assigned "correction factor" for managing hyperglycemia.
3. Age 18-75 years, inclusive.
4. Random serum C-peptide concentration < 0.5 ng/mL.
5. Willingness to follow all study procedures, including attending all clinic visits.
6. Subject has provided informed consent as evidenced by a signed/dated informed consent form completed before any trial-related activities occur.

Exclusion Criteria:

1. Pregnancy: For women of childbearing potential, there is a requirement for a negative urine pregnancy test and for agreement to use contraception throughout the study and for 7 days after the last dose of study glucagon. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
2. Breastfeeding: Nursing mothers will be allowed into the study. However, breast feeding during the during inpatient study visits and for 48 hours after each dose of study drug is not allowed.
3. HbA1c >9.0% at Screening.
4. BMI > 40 kg/m2.
5. Renal insufficiency (serum creatinine greater than 3.0 mg/dL) or end-stage renal disease. requiring renal replacement therapy.
6. Serum ALT or AST equal to or greater than 3 times the upper limit of normal.
7. Hepatic synthetic insufficiency as defined as a serum albumin of less than 3.0 g/dL.
8. Hematocrit of less than or equal to 30%.
9. BP readings at Screening where SBP <90 or >150 mm Hg, and DBP <50 or >100 mm Hg.
10. Clinically significant ECG abnormalities.
11. Use of > 2.0 U/kg total insulin dose per day.
12. Inadequate venous access.
13. Congestive heart failure, NYHA class III or IV.
14. History of myocardial infarction, unstable angina, or revascularization within the past 6 months.
15. History of a cerebrovascular accident in past 6 months or with major neurological deficits.
16. Active malignancy within 5 years from Screening, except basal cell or squamous cell skin cancers. History of breast cancer or malignant melanoma will be exclusionary.
17. Major surgical operation within 30 days prior to Screening.
18. Current seizure disorder (other than with suspect or documented hypoglycemia).
19. Current bleeding disorder, treatment with warfarin, or platelet count below 50 x 10e9 per liter.
20. History of pheochromocytoma or disorder with increased risk of pheochromocytoma (MEN 2, neurofibromatosis, or Von Hippel-Lindau disease).
21. History of insulinoma.
22. History of allergies to glucagon or glucagon-like products, or any history of significant hypersensitivity to glucagon or any related products or to any of the excipients (DMSO & trehalose) in the investigational formulation.
23. History of glycogen storage disease.
24. Subject tests positive for HIV, HCV or HBV infection (HBsAg+) at Screening.
25. Active substance or alcohol abuse (more than 21 drinks/wk. for males or 14 drinks/wk. for females). Subjects reporting active marijuana use or testing positive for tetrahydrocannabinol (THC) via rapid urine test will be allowed to participate in the study at the discretion of the Investigator.
26. Administration of glucagon within 28 days of Screening.
27. Participation in other studies involving administration of an investigational drug or device within 30 days or 5 half-lives, whichever is longer, before Screening for the current study and during participation in the current study.
28. Any reason the Investigator deems exclusionary.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - ProSciento, Inc., Chula Vista, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rainier Clinical Research Center, Inc., Renton, Washington
- Canada (2):
  - LMC ESD, Inc., Toronto, Ontario
  - Altasciences Algorithme Pharma, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christiansen MP, Cummins M, Prestrelski S, Close NC, Nguyen A, Junaidi K. Comparison of a ready-to-use liquid glucagon injection administered by autoinjector to glucagon emergency kit for the symptomatic relief of severe hypoglycemia: two randomized crossover non-inferiority studies. BMJ Open Diabetes Res Care. 2021 Oct;9(1):e002137. doi: 10.1136/bmjdrc-2021-002137. PMID 34620618

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period began 08 Jan 2018 and ran through 02 Apr 2018. Subjects were screened for study eligibility at one of the six clinical sites up to 30 days prior to randomization.
Pre-assignment Details: A total of 81 eligible subjects were randomized to treatment. However, two subjects withdrew consent prior to dosing, so the number of subjects exposed to study treatment was 79.
Period: Overall Study
Arm/Group | G-Pen Followed by Lilly Glucagon | Lilly Glucagon Followed by G-Pen
Started | 41 | 40
Completed | 39 (1 subject dropped before G-Pen; another after G-Pen (n=40 G-Pen; N=39 Lilly Glucagon)) | 36 (1 subject dropped before Lilly Glucagon; 3 others after Lilly Glucagon (N=39 Lilly; N=36 G-Pen))
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- All Randomized Subjects: A total of 81 subjects met eligibility requirements and were randomized to study treatment.
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 71
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  North America | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Positive Glucose Response
Description: Increase in plasma glucose concentration from below 50.0 mg/dL to greater than 70.0 mg/dL within 30 minutes after receiving glucagon
Time Frame: 0 to 30 minutes post dose
Population: Intent to treat analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
Participants | 76 | 78

2. Secondary Outcome: Time for Positive Glucose Response
Description: Time from administration of glucagon for plasma glucose to rise from below 50.0 mg/dL to above 70.0 mg/dL
Time Frame: 0 to 180 minutes post dose
Population: Intent-to treat analysis population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
minutes | 12.17 (3.604) | 8.58 (2.026)

3. Secondary Outcome: Number of Subjects With a Positive Response for the Combination Endpoint: Positive Glucose Response/Positive Glucose Increase
Description: A positive response for this endpoint is a return of plasma glucose to > 70 mg/dL or an increase in plasma glucose by ≥20 mg/dL within 30 minutes after receiving glucagon
Time Frame: 0 to 30 minutes post dose
Population: Intent to treat analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
Participants | 76 | 78

4. Secondary Outcome: Number of Subjects With a Positive Glucose Increase
Description: Increase in plasma glucose by ≥ 20.0 mg/dL within 30 minutes after receiving glucagon
Time Frame: 0 to 30 minutes post dose
Population: Intent to treat analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
Participants | 76 | 78

5. Secondary Outcome: Time for Positive Glucose Increase
Description: Time from administration of glucagon for plasma glucose to increase by ≥20 mg/dL from baseline
Time Frame: 0 to 180 minutes post dose
Population: Intent to treat analysis population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
minutes | 11.36 (3.345) | 8.02 (1.856)

6. Secondary Outcome: Number of Subjects With a Positive Response for the Combination Endpoint: Positive Glucose Response/Relief of Neuroglycopenic Symptoms
Description: A positive response for this endpoint is a return of plasma glucose to > 70 mg/dL or clearance of all neuroglycopenic symptoms of hypoglycemia within 30 minutes after receiving glucagon. Four symptoms were assessed: dizziness, blurred vision, difficulty in thinking and faintness.
Time Frame: 0 to 30 minutes post dose
Population: Intent to treat analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
Participants | 76 | 78

7. Secondary Outcome: Number of Subjects With Relief of Neuroglycopenic Symptoms
Description: Clearance of all neuroglycopenic symptoms of hypoglycemia within 30 minutes after receiving glucagon. Four symptoms were assessed: dizziness, blurred vision, difficulty in thinking and faintness.
Time Frame: 0 to 30 minutes post dose
Population: Intent to treat analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
Participants | 74 | 77

8. Secondary Outcome: Time to Resolution of Autonomic Symptoms
Description: Time from administration of glucagon to complete resolution of 4 autonomic symptoms of hypoglycemia. Symptoms included: sweating, tremor, palpitations and feeling of nervousness.
Time Frame: 0 to 180 minutes post dose
Population: Intent to treat analysis population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
minutes | 13.8 (10.89) | 12.0 (7.44)

9. Secondary Outcome: Time to Resolution of Neuroglycopenic Symptoms
Description: Time from administration of glucagon to complete resolution of 4 neuroglycopenic symptoms of hypoglycemia. Four symptoms were assessed: dizziness, blurred vision, difficulty in thinking and faintness.
Time Frame: 0 to 180 minutes post dose
Population: Intent to treat analysis population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
minutes | 14.2 (15.12) | 12.2 (8.85)

10. Secondary Outcome: Time to Resolution of the Feeling of Hypoglycemia
Description: Time from administration of glucagon to resolution of the overall sensation of hypoglycemia. Subjects were asked to answer yes/no to the question, "Do you feel hypoglycemic?" The time point as which the subject first answered "no" was considered the time of resolution.
Time Frame: 0 to 180 minutes post dose
Population: Intent to treat analysis population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
minutes | 11.6 (6.45) | 13.1 (7.86)

11. Secondary Outcome: Glucose AUC
Description: Area under the curve for plasma glucose.
Time Frame: 0 to 180 minutes post dose - Blood samples for assessment of blood glucose concentration were collected every 5 minutes post-dose to 90 minutes, and then at 120, 150 and 180 minutes post dose.
Population: Intent to treat analysis population. Due to missing data AUC was only evaluable in 67 subjects per arm.
Measure: Mean (Standard Deviation); unit: mg∙min/dL
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 67 | 67
mg∙min/dL | 33686.04 (5300.204) | 33538.60 (5705.219)

12. Secondary Outcome: Glucose Cmax
Description: Maximum concentration of plasma glucose.
Time Frame: as for outcome 11
Population: Intent to treat analysis population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
mg/dL | 238.32 (45.626) | 228.11 (46.567)

13. Secondary Outcome: Glucose Tmax
Description: Time to maximum concentration of plasma glucose. Blood samples for assessment of blood glucose concentration were collected every 5 minutes post-dose to 90 minutes, and then at 120, 150 and 180 minutes post dose.
Time Frame: 0 to 180 minutes post dose
Population: Intent to treat analysis population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
minutes | 125.67 (33.513) | 113.89 (31.908)

14. Secondary Outcome: Glucagon Preparation and Administration Time
Description: Time required to prepare and inject glucagon as measured between a "decision to dose" and completion of the injection
Time Frame: 0 to 5 minutes pre-dose
Population: Intent to treat analysis population
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 78
seconds | 27.3 (19.66) | 97.2 (45.06)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 9 weeks, from the time of consent through the follow-up visit.
Description: Treatment-Emergent Adverse Events
  Note: Some subjects experienced multiple adverse events. Consequently, the sum of the number of subjects experiencing each individual adverse events is greater than the number of unique subjects experiencing at least one adverse event.
Groups:
- G-Pen: G-Pen: 1 mg subcutaneous injection of G-Pen (glucagon injection) administered via auto-injector. Between the 2 arms, a total of 76 subjects received a dose of G-Pen in the study.
- Lilly Glucagon: Lilly Glucagon: 1 mg subcutaneous injection of Lilly Glucagon (glucagon injection [RNDA Origin]). Between the 2 arms, a total of 78 subjects received a dose of Lilly Glucagon in the study.
Arm/Group | G-Pen | Lilly Glucagon
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/78
Other Adverse Events (participants affected / at risk) | 46/76 | 34/78
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | G-Pen (N=76) | Lilly Glucagon (N=78)
Headache (Nervous system disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 29 | 26
Vomiting (Gastrointestinal disorders) | 20 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the Institution nor the principal investigator may submit for publication or presentation, the results of this trial without prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT03439072/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT03439072/SAP_001.pdf